CLINICAL TRIAL: NCT07165340
Title: Evaluation of Lymphatic Response to Treatment in Patients With Edema Secondary to Superficial Venous Disease
Brief Title: Evaluation of Lymphatic Response to Physiotherapy in Patients With Swelling Associated With Superficial Venous Disease
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Tactile Medical (Industry)
Responsible Party: Principal Investigator, John Rasmussen, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-25-0191
Record Dates: First submitted 2025-08-19; First posted 2025-09-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Venous Disease
Keywords: near-infrared fluorescence lymphatic imaging; lymphatic imaging; pneumatic compression therapy; indocyanine green; chronic venous disease
MeSH Terms: interventions — Ultrasonography, Doppler, Duplex; Compression Bandages

STUDY DESIGN:
Intervention Model Description: This is a blinded, prospective, 2-arm, randomized study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control Arm (Active Comparator): Subjects will receive standard-of-care compression bandaging.
  Interventions: Combination Product: Indocyanine Green near infrared fluorescence imaging; Diagnostic Test: Duplex ultrasound; Device: compression wrap
- Treatment Arm (Experimental): Subjects will receive both standard-of-care compression bandaging AND daily treatments with an advanced pneumatic compression device.
  Interventions: Combination Product: Indocyanine Green near infrared fluorescence imaging; Device: advanced pneumatic compression; Diagnostic Test: Duplex ultrasound; Device: compression wrap

INTERVENTIONS:
Combination Product: Indocyanine Green near infrared fluorescence imaging — A total of 10 intradermal injections of 25 ug indocyanine green (ICG) in 0.1 mL saline are administered in the feet, medial ankles, lateral calves, and thigh. The total dose of ICG will not exceed 250 ug. After injection, the legs will be illuminated by the dim output of a 780 nm laser diode, and the resultant fluorescent signal emanating from ICG-laden lymph will be collected by a custom built near-infrared fluorescent lymphatic imager.
  Other Names: near-infrared fluorescence lymphatic imaging
Device: advanced pneumatic compression — The advanced pneumatic compression device (APCD) mimics manual lymphatic drainage, a light massage that stimulates lymphatic uptake and function and frequently prescribed for lymphedema therapy. Daily treatment will be prescribed for approximately 30 days.
  Arms: Treatment Arm
Diagnostic Test: Duplex ultrasound — Duplex ultrasound to measure venous reflux will be done at each visit.
Device: compression wrap — A compression wrap, to provide 20-40 mm Hg of pressure, will be provided for daily use between visits (approximately 30 days).

SUMMARY:
This study seeks to demonstrate the effect of advanced pneumatic compression in treatment naïve patients with CEAP C3 and C4 chronic venous disease. The main questions it aims to answer are:

* Does lymphatic treatment improve lymphatic function following ~30 days of advanced pneumatic compression device therapy?
* Does lymphatic dysfunction correlate with CEAP score and venous reflux times? Over the course of 30-45 days, participants will undergo two sessions of near-infrared fluorescence lymphatic imaging to assess whether advanced pneumatic compression treatment improves lymphatic (dys)function. Subjects will be divided into two groups, a treated and a control group. Both groups will receive standard-of-care compression bandaging. The treated group will also be asked to complete daily sessions of pneumatic compression therapy at home. At both imaging sessions, duplex ultrasound will also be used to assess venous reflux times. Researchers will compare the changes in lymphatic and venous (dys)function between the two groups to see if lymphatic function improves with pneumatic compression treatment and if they dysfunction is correlated with CEAP clinical score and venous reflux times.

ELIGIBILITY:
Inclusion Criteria:

1. Participant >18 years of age
2. Participant with an objective diagnosis of CEAP Class 3 or 4 superficial venous disease (superficial reflux time >0.5 sec), with venous edema (revised VCSS score of 2 or 3 for edema).
3. Participant must provide informed consent
4. Participant is willing and able to fulfill study timeline
5. Participant is a candidate for APCD treatment per the FTP indications
6. Lymphatic dysfunction is observed, using NIRF-LI, in affected limb.

Exclusion Criteria:

1. History of pelvic or lower extremity cancers
2. Systemic organ failure including heart failure
3. BMI >35
4. Previous endovascular or open vascular interventions
5. Patients with known, or family history of, primary lymphedema
6. Prior use of advanced pneumatic compression device, or complete decongestive therapy (CDT) on the lower extremities
7. Peripheral arterial disease with ABI <0.8
8. Participants with deep venous obstruction
9. Skin disease not related to CVD
10. Participants with iodine allergies including patients with shellfish allergy who may be allergic to iodine that may be in the ICG formulation
11. Females who are pregnant or breastfeeding
12. Females with the intent of becoming pregnant within 30 days after participation in final imaging session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Extent of Dermal Backflow | Assessed at Visit 1 and 2 (approximately 30 days apart)
  The area of abnormal dermal lymphatic backflow in the leg.
Lymphatic pumping rate | Assessed at Visit 1 and Visit 2 (approximately 30 days apart)
  Number of pumping events observed per minute assessed in the medial ankle.

SECONDARY OUTCOMES:
Correlation of CEAP score and lymphatic pumping rates | Assessed at Visit 1 and 2 (approximately 30 days apart)
Correlation of CEAP score with extent of dermal backflow | Assessed at Visit 1 and 2 (approximately 30 days apart)
Change in limb volume between arms. | Assessed at Visit 1 and 2 (approximately 30 days apart)
  Limb volume, determined from limb circumference measurements, will be assessed at both visits.
Change in LLIS score between arms | Assessed at Visit 1 and 2 (approximately 30 days apart)
  Patient reported outcomes assessed using the Lymphedema Life Impact Scale (LLIS) at each visit and change determined after Visit 2. Possible scores range from 0 to 100 with a higher score indicating a greater impact of disease on quality of life.
Change in Venous Clinical Severity Score (VCSS) between arms | Assessed at Visit 1 and 2 (approximately 30 days apart)
  Venous Clinical Severity Score (VCSS) will be assessed at each visit. Possible scores range from 0 to 30 with a higher score indicating a greater severity of vascular disease.
Change in patient reported outcomes between arms | Assessed at Visit 1 and 2 (approximately 30 days apart)
  Patient reported outcomes assessed using the Lower Extremity Functional Scale (LEFS) at each visit and change determined after Visit 2. Possible scores range from 0 to 80 with a higher score indicating a greater impact of disease on limb functionality.

CONTACTS AND LOCATIONS:
Overall Officials: John C Rasmussen, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston/UTPhysicians, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published in a scientific journal along with description of protocol. The complete data set includes large (GBs) sequences of images that may include protected health information (tattoos). Partial, redacted data sets may be sharable upon request.